CLINICAL TRIAL: NCT06055517
Title: A Phase-2 Trial to Investigate the Use of Pulsed Low-dose Rate Re-irradiation for Recurrent Glioma (PULSAR)
Brief Title: Use of Pulsed Low-dose Rate Re-irradiation for Recurrent Glioma (PULSAR)
Acronym: PULSAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO-2022-82
Record Dates: First submitted 2023-09-13; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Heart Rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulsed low dose-rate radiotherapy (pLDRT) (Experimental)
  Interventions: Radiation: Pulsed low dose-rate radiotherapy (pLDRT)

INTERVENTIONS:
Radiation: Pulsed low dose-rate radiotherapy (pLDRT) — Radiation treatment will be carried out with high-energy photons (6MV) using intensity modulated radiation therapy (IMRT) or volumetric arc radiation therapy (VMAT). The daily dose is 2 Gy, divided into 10 subfractions of 0.2 Gy spaced by 3 minutes. The cumulative dose will be individualized for each patient and can range from a minimum of 40 Gy to a maximum of 60 Gy.

SUMMARY:
Re-irradiation in gliomas is a therapeutic option at recurrence before of 2nd-line chemotherapy. The dose of re-irradiation with conventional fractionation is unfortunately limited by the risk of symptomatic radionecrosis that is significant for cumulative doses above 100 Gy. The use of unconventional low dose rate pulsed radiotherapy (pLDRT) can reduce the risk of radiotoxicity while taking advantage of the cellular hyper-radiosensitivity that occurs at low dose-rates. The present study therefore aims at evaluating whether the use of pLDRT in the re-irradiation of recurrences of gliomas allows maintaining a low risk of symptomatic radionecrosis even for cumulative doses greater than 100 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Ability to express appropriate informed consent to treatment;
* Diagnosis of cerebral glioma;
* Histological/radiological confirmation of disease recurrence/relapse;
* Previous brain-level radiation therapy completed a minimum of 6 months;
* Performance status: ECOG=0-2.

Exclusion Criteria:

* Refusal to radiation treatment (i.e., absence of informed consent signed);
* Concomitant chemotherapy;
* Leptomeningeal spread of disease and localization in both cerebral hemispheres;
* Current pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2028-05-26 (Estimated); Study Completion 2028-05-26 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of brain radionecrosis in patients undergoing re-irradiation of brain tumors with pulsed low-dose-rate schedule | up to 5 years
  Incidence of grade >=2 brain radionecrosis in patients undergoing re-irradiation of brain tumors with pulsed low-dose-rate schedule, defined according to CTCAE v5.0 scale

SECONDARY OUTCOMES:
To assess the median time to local disease progression | up to 5 years
  Assessment of median disease progression-free survival. PFS will be defined as the time from study enrollment until progression or death for any cause, whichever comes first. Disease progression defined according to RANO criteria.
To assess the median survival time | up to 5 years
  Assessment of median survival time. Survival will be defined as the time from study enrollment until death for any cause
To assess the incidence of toxicities other than radionecrosis | up to 5 years
  Assessment of incidence of other neurological toxicities graded with the scale CTCAE v 5.0
To assess the presence of biomarkers associated with the actinic toxicity | up to 5 years
  Frequency of selected circulating biomarkers in patients with actinic toxicity
To assess the presence of biomarkers associated with response to therapy | up to 5 years
  Difference in progression free survival (PFS) probability between groups of patients with or without selected circulating biomarkers. PFS will be defined as the time from study enrollment until progression or death for any cause, whichever comes first. Median survival for each biomarker will be calculated
To assess the presence of biomarkers associated with overall survival (OS) | up to 5 years
  Difference in OS probability between groups of patients with or without selected circulating biomarkers. OS will be defined as the time from study enrollment until death for any cause
To evaluate the immunomodulation induced by the pulsed schedule in comparison with the conventional schedule | up to 5 years
  Difference in the frequency of immunotherapeuthic markers between pulsed and conventional radiotherapy schedules

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Vinante, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO); Lorena Baboci, PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO)
Locations (1):
- IRCCS-Centro di Riferimento Oncologico (CRO) di Aviano, Aviano, Pordenone, Italy